CLINICAL TRIAL: NCT06705400
Title: The Bloom Study - a Safe and Healthy Start in Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: National Institute of Public Health, University of Southern Denmark (Unknown); Danish Centre for Health Economics (DaCHE), University of Southern Denmark (Unknown); University of Copenhagen (Other); Danish Research Centre for Migration, Ethnicity and Health, University of Copenhagen (Unknown); Centre for Childhood Health (Unknown); The Centre for Health Economics, University of York (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-24032126
Record Dates: First submitted 2024-11-14; First posted 2024-11-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Overweight, Childhood; Obesity in Children
Keywords: The Bloom Study; Intervention; Infants; Weight status; Community health nurses; Home-based; Randomized controlled trial; Children; Multi-component; Health promotion and prevention; Overweight; Obesity; Food habits and meals; Motor skills and movement; Screen use; Sleep
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Feeding Behavior | interventions — Movement; Sleep; Food; Meals

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Bloom Intervention adds to standard municipal care (5-6 home visits) with a prenatal visit, visits at 18 and 30 months, up to eight phone consultations, parent groups, and a video library.
  Home visits: Three extra visits include one in pregnancy week 22-24 to build trust and assess needs using a dialogue tool focused on social and demographic factors. Visits at 18 and 30 months support sustained progress and address new challenges.
  Phone consultations: Up to eight calls support breastfeeding, bottle-feeding, and complementary feeding. Phone consultations at 12 and 24 months aid in maintaining healthy habits during key transitions, like starting daycare.
  Parent groups: Encourage shared experiences among parents, with policies promoting father participation.
  Video library: Includes 62 videos on nutrition, motor skills, sleep, etc., with 48 available in multiple languages for wider access.
  Interventions: Behavioral: Multi-behavioural
- Control (No Intervention): The families in the control municipalities will receive standard deliveries from the community health nurses

INTERVENTIONS:
Behavioral: Multi-behavioural — The Bloom Study is implemented in an existing and highly accepted health service delivered by community health nurses. Beyond focusing on food, meals, motor skills and movement, the intervention also target sleep and family sense of security. The intervention commence in pregnancy and continues until the child is 2½ years old.
  Other Names: Motor skills and movement; Screen use; Sleep; Family sense of security; Food and meals
  Arms: Intervention

SUMMARY:
The aim of the Bloom Study is to promote healthy weight development among infants through a home-based health promoting intervention implemented in the Danish setting of community health nurses. The intervention begins during pregnancy and runs until the child reaches the age of 30 months.

The Bloom Intervention was developed over a six-year period from 2017 to 2023 according to the Intervention Mapping approach and based on a co-creation process.

The Bloom Intervention is evaluated in a cluster-randomized trial involving 22 Danish municipalities (11 intervention and 11 control). All children born from first-time mothers over a period of 12 months are invited to participate.

DETAILED DESCRIPTION:
Childhood overweight and obesity are major public health challenges. In Denmark, 14% of children have overweight or obesity at school entry, rising to 19% by school leaving, with higher prevalence levels among children from low socio-economic positions and ethnic minority backgrounds.

Early intervention is crucial since childhood obesity is hard to reverse, and infancy presents an opportunity to address modifiable risk factors. It is well-documented that both genetic, behavioral, psychosocial, and environmental factors play key roles. Modifiable risk factors include feeding practices, physical activity, screen use, and sleep. Additionally, growing evidence suggests that psychological stress in early life due to unmet socio-emotional needs may lead to disrupted energy balance homeostasis, resulting in weight gain.

The Bloom Study is designed to address food and meals, motor skills and movement, screen use, sleep, and sense of security in the family. The intervention targets first-time families, with a special focus on reaching all families across varying socio-economic positions and ethnic backgrounds. Also, the Bloom intervention has a strong focus on involving fathers/partners. It is delivered through the established and highly accepted system of community health nurses in Denmark.

The intervention is initiated during pregnancy and continues until the child reaches 30 months of age. The main intervention components include: 1) an extra home visit during pregnancy, 2) an extra home visit when the child ais 18 months, 3) an extra home visit when the child is 30 months, 3) telephone consultations, 4) parent groups, and 5) a video library for parents.

An important element of the implementation strategy is to ensure that the intervention design and implementation are compatible with the existing practices, priorities, and values within the system of Danish community health nurses. Additionally, the implementation of the Bloom Study will be supported by five main activity components: 1) training of community health nurses including a five-day training course, supervision, and a comprehensive implementation manual containing instructions for standardized delivery of the intervention, 2) selection of local program ambassadors among community health nurses in the municipalities, 3) regular contact with the research group including assignment of one main contact person, 4) meeting activities including start-up meetings, network meetings across municipalities, and local staff meetings, and 5) partial economic compensation.

The Bloom Study is evaluated within a cluster-randomized controlled trial (cluster-RCT) with 22 municipalities randomly allocated to intervention (11 municipalities) and control (11 municipalities). The intervention is initiated during pregnancy and continues until the child reaches 30 months of age. Follow-up data are collected at child age of 36 months. Primary outcome is Body Mass Index (BMI) z-score at child age of 36 months.

ELIGIBILITY:
Inclusion Criteria:

All children born from first-time mothers being in gestation week 20 between November 1st 2024 and October 31st 2025.

Exclusion Criteria:

Not being able to receive digital post.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3500 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
BMI z-score | 36 months
  Between group difference in BMI z-score based on WHO references. Weight is measured by portable weights (Seca 887) and height is measured by measurement tapes according to a standardized instruction.

SECONDARY OUTCOMES:
Weight status | 36 months
  Between group difference in prevalence of children with underweight, overweight and obesity based on WHO references. Weight is measured by portable weights (Seca 887) and height is measured by measurement tapes according to a standardized instruction.
BMI z-score | Few days after birth, Within first week after returning to home, Within first months, 2 months, 4-6 months, 8-10 months, 18 months, 30 months
  Between group difference in BMI z-score based on WHO references.
  From birth to 10 months weight is measured by portable weights approved for standard use by community health nurses and according to a standardized instruction (journal records).
  At age 18 and 30 months, weight is measured by portable weights (Seca 887).
  From birth to 18 months length is measured by a mobile measuring mat (Seca 201) according to a standardized instruction.
  At age 30 months, height is measured by measurement tapes according to a standardized instruction.
Fat mass (kg) | 36 months
  Between group difference in fat mass measured by bioimpedance analysis. Bioimpedance will be measured by the Impedimed SFB7 device.
Fat free mass (kg) | 36 months
  Between group difference in fat free mass measured by bioimpedance analysis. Bioimpedance will be measured by the Impedimed SFB7 device.
Fat mass index in kg/m2 | 36 months
  Between group difference in fat mass index measured by bioimpedance analysis. Bioimpedance will be measured by the Impedimed SFB7 device.
Fat free mass index (kg/m2) | 36 months
  Between group difference in fat free mass index measured by bioimpedance analysis. Bioimpedance will be measured by the Impedimed SFB7 device.
% Fat mass | 36 months
  Between group difference in % fat mass index measured by bioimpedance analysis. Bioimpedance will be measured by the Impedimed SFB7 device.
% Fat free mass | 36 months
  Between group difference in % fat free mass index measured by bioimpedance analysis. Bioimpedance will be measured by the Impedimed SFB7 device.

OTHER OUTCOMES:
Child social-emotional development | 12, 24 and 36 months
  Measurement instrument: The Ages & Stages Questionnaires: Social-Emotional, Second Edition (ASQ:SE-2) (parents' questionnaires). The questionnaire includes a total of 27 (12 months), 31 (24 months) and 36 (36 months) questions each with possible scores of 0, 5, 10 or 15 from which a total sum score is generated. A higher score indicates a higher extent of socio-emotional concerns.
Child mental health | 24 and 36 months
  Measurement instrument: Strengths and Difficulties Questionnaire (SDQ, 2-4 years) (parents' questionnaires) The instrument five subscales: Conduct problems (score range from 0-10); emotional symptoms (score range from 0-10); hyperactivity (score range from 0-10); peer problems (score range from 0-10); and prosocial behaviour (score range from 0-10). A total difficulties score can be generated by summing the scores of all scales except the prosocial behaviour scale (score range from 0-40). The extent of difficulties increases with increasing score.
Child eating behaviour | 24 and 36 months
  Measurement instrument: Child Eating Behaviour Questionnaire (BEBH) (parents' questionnaires) The questionnaire covers eight domains: Food responsiveness, Emotional over-eating, Enjoyment of food, Desire to drink, Satiety responsiveness, Slowness in eating, Emotional under-eating and Food fussiness.
  For each item the response categories (including scoring) is: Never=1, Rarely=2, Sometimes=3, Often=4, Always=5, from which a domain mean score is generated. Higher scores indicate more frequent demonstrations of behaviours characterizing the trait of the domain.
Parental feeding practices - < 2 years, milk | 6 months
  Measurement instrument: The Feeding Practices and Structure Questionnaire (< 2 years, milk) The complete measure comprises a total of 18 items, scored on a 5-point Likert scale with higher scores indicating greater endorsement of that practice.
  The complete questionnaire covers four domains of non-responsive feeding practices. The following two domains are included at 6 months: Using food to calm (5 items), and Parent-led feeding (6 items).
Parental feeding practices - < 2 years, solid food | 12 months
  Measurement instrument: The Feeding Practices and Structure Questionnaire (< 2 years, solid food) The measure comprises a total of 34 items, scored on a 5-point Likert scale with higher scores indicating greater endorsement of that practice.
  The questionnaire covers six domains of non-responsive feeding practices: Feeding on demand (4 items), Using food to calm (6 items), Persuasive Feeding (7 items), Parent-led feeding (4 items), Family meal environment (4 items), and Using (non-) food rewards (9 items).
Parental feeding practices, >= 2 years | 24 and 36 months
  Measurement instrument: The Feeding Practices and Structure Questionnaire (FPFQ-28) The measure comprises a total of 28 items, scored on a 5-point Likert scale with higher scores indicating greater endorsement of that practice.
  The questionnaire covers seven domains of non-responsive feeding practices: Reward for Behaviour (4 items), Reward for Eating (4 items), Persuasive Feeding (6 items), Overt Restriction (4 items), Covert Restriction (4 items), Structured Meal Setting (3 items), and Structured Meal Timing (3 items).
Parents' self-efficacy related to child sleep | 6, 12, 24 and 36 months
  Measurement instrument: Uppsala Parental Self-Efficacy about Infant Sleep Instrument (UPPSEISI)(parents' questionnaires) The UPPSEISI includes 11 items with total scores ranging from 11 to 55 points. Higher values on UPPSEISI indicate a higher level of parental self-efficacy. The 11 items cover two domains: The Child's Need for Sleep (CNS) domain (8 items), and the Arduous Parenting (AP) domain (3 items).
Parents' well-being | 6, 12, 24 and 36 months
  Measurement instrument: WHO5 (parents' questionnaires) The WHO-5 index is scored based on responses to five statements rated on a 6-point Likert scale.
  The raw sum score ranges from 0 to 25. Higher scores indicate better well-being.
Parents' self-efficacy related to parenthood | 6, 12, 24 and 36 months
  Measurement instrument: Perceived Maternal Parenting Self-Efficacy (PMP S-E) tool (parents' questionnaires). The complete tool consists of 20 items. Higher scores indicate higher self-efficacy.
  The complete tool covers four domains. The following domain is included: Evoking behaviour (7 items).
Parental stress | 6, 12, 24 and 36 months
  Measurement instrument: The 16-item version of the Parental Stress Scale (parents' questionnaires) (Pontoppidan et al., 2018). The scale applies a five-point response key. Overall possible scores on the scale range from 16 - 80. The higher the score, the higher the measured level of parental stress.
Sensitive parenting | 6, 12, 24 and 36 months
  Measurement instrument: The Parental Reflective Functioning Questionnaire (PRFQ), subscale Certainty about Mental States (parents' questionnaires)
  The subscale includes 6 items with a seven-point response key. The higher the mean score, the higher the degree of sensitive parenting.
Breastfeeding | 6, 12 and 24 months
  Indicators: 1) Ever breastfeeding, 2) Duration of exclusive breastfeeding, 3) Duration of partial breastfeeding.
  Measurement tool: Developed for the study
Bottle feeding with infant milk formula | 6 and 24 months
  Indicators: 1) Ever given infant milk formula, 2) Amount of daily infant milk formula at 6 months of age, 3) Duration of bottle feeding (infant milk formula) Measurement tool: Developed for the study
Introduction to complementary food | 6 and 12 months
  Indicator: Age (in months and weeks) at introduction to complementary food Measurement tool: Developed for the study
Use of baby food squeeze pouches | 6 and 12 months
  Indicators: 1) Ever use of baby food squeeze pouches, 2) Method for feeding the child from the food squeeze pouch Measurement tool: Developed for the study
Child screen use | 6, 12, 24 and 36 months
  Indicators: 1) Daily screen watching time, 2) Frequency of screen use for soothing Measurement tool: Developed for the study
Child sleep | 6, 12, 24 and 36 months
  Indictors: 1) Child night-time sleep duration and 2) Child night-time sleep quality Measurement tool: Developed for the study
Motor skills | 6 months
  Indicator: Frequency of tummy time Measurement tool: Developed for the study
Movement | 6 and 12 months
  Indicator: Frequency of active play with the child Measurement tool: Developed for the study
Child placed in fixed sedentary position | 6 and 12 months
  Indicator: Time (daily) child fixed in sedentary sitting position Measurement tool: Developed for the study

CONTACTS AND LOCATIONS:
Overall Officials: Camilla T Bonnesen, Principal Investigator — National Institute of Public Health, University of Southern Denmark
Locations (1):
- National Institute of Public Health, University of Southern Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Access Criteria: A formal application with reasonable request must be approved by the study's management group. Data will only be shared as long as there is a legal basis for the disclosure.

REFERENCES:
- [Derived] Bonnesen CT, Rasmussen M, Kierkegaard L, Carlsson RR, Jensen MP, Ubbesen TR, Madsen KR, Thygesen LC, Krolner RF, Brautsch LAS, Rosing JA, Kongstad LP, Vaever MS, Egmose I, Pedersen TP. Study protocol for a cluster-randomized controlled trial of a universal home-based, multi-component intervention to promote healthy weight development in children during infancy and toddlerhood in denmark: the bloom study. BMC Public Health. 2025 Aug 27;25(1):2952. doi: 10.1186/s12889-025-24352-1. PMID 40866846
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/40866846/
- Available data/document: Statistical Analysis Plan — https://findresearcher.sdu.dk/ws/portalfiles/portal/298847036/Statistical_Analysis_Plan_for_the_Bloom_Study_14112025_FINAL.pdf